CLINICAL TRIAL: NCT05933187
Title: A Phase 1, Open-label Trial to Evaluate the Pharmacokinetics and Relative Bioavailability of Emraclidine Following a Single Oral Administration of Immediate-Release Tablets in Healthy Adult Participants
Brief Title: A Study Evaluating the Pharmacokinetics and Relative Bioavailability of Emraclidine Immediate-Release Tablets in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CVL-231-HV-1013
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Intervention Model Description: This is a 4-period, 4-sequence crossover study. The 4 treatments are A- 30 milligrams (mg) emraclidine IR tablets (reference); B- 30 mg emraclidine IR test tablets 1; C- 30 mg emraclidine IR test tablets 2; D- 30 mg emraclidine IR test tablets 3. Participants will be randomized to 1 of 4 treatment sequences. Each participant will be administered each of the 4 treatments exactly once, i.e.,1 treatment per period and there will be a 7 day washout period between each treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1: A-B-C-D (Experimental): Participants will receive emraclidine, 30 mg IR tablets, in the treatment sequence A-B-C-D orally, on Day 1 of each 5-day treatment period (up to 26 days)
  Interventions: Drug: Treatment A: Emraclidine 30mg IR tablets (reference); Drug: Treatment B: Emraclidine 30mg IR test tablets 1; Drug: Treatment C: Emraclidine 30mg IR test tablets 2; Drug: Treatment D: Emraclidine 30mg IR test tablets 3
- Sequence 2: B-C-D-A (Experimental): Participants will receive emraclidine, 30 mg IR tablets, in the treatment sequence B-C-D-A orally, on Day 1 of each 5-day treatment period (up to 26 days)
  Interventions: Drug: Treatment A: Emraclidine 30mg IR tablets (reference); Drug: Treatment B: Emraclidine 30mg IR test tablets 1; Drug: Treatment C: Emraclidine 30mg IR test tablets 2; Drug: Treatment D: Emraclidine 30mg IR test tablets 3
- Sequence 3: C-D-A-B (Experimental): Participants will receive emraclidine, 30 mg IR tablets, in the treatment sequence C-D-A-B orally, on Day 1 of each 5-day treatment period (up to 26 days)
  Interventions: Drug: Treatment A: Emraclidine 30mg IR tablets (reference); Drug: Treatment B: Emraclidine 30mg IR test tablets 1; Drug: Treatment C: Emraclidine 30mg IR test tablets 2; Drug: Treatment D: Emraclidine 30mg IR test tablets 3
- Sequence 4: D-A-B-C (Experimental): Participants will receive emraclidine, 30 mg IR tablets, in the treatment sequence D-A-B-C orally, on Day 1 of each 5-day treatment period (up to 26 days)
  Interventions: Drug: Treatment A: Emraclidine 30mg IR tablets (reference); Drug: Treatment B: Emraclidine 30mg IR test tablets 1; Drug: Treatment C: Emraclidine 30mg IR test tablets 2; Drug: Treatment D: Emraclidine 30mg IR test tablets 3

INTERVENTIONS:
Drug: Treatment A: Emraclidine 30mg IR tablets (reference) — IR oral tablets
  Other Names: CVL-231
Drug: Treatment B: Emraclidine 30mg IR test tablets 1 — IR oral tablets
  Other Names: CVL-231
Drug: Treatment C: Emraclidine 30mg IR test tablets 2 — IR oral tablets
  Other Names: CVL-231
Drug: Treatment D: Emraclidine 30mg IR test tablets 3 — IR oral tablets
  Other Names: CVL-231

SUMMARY:
The purpose of this trial is to evaluate plasma concentrations of emraclidine following single dose oral administration of different emraclidine immediate release (IR) tablets in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women of childbearing potential must agree to use at least an acceptable birth control method, during the trial and for 7 days after the last dose of investigational medicinal product (IMP)
* Body mass index of 18.5 to 35.0 kilogram/meter square (kg/m^2), inclusive, and a total body weight ≥50 kg
* Healthy as determined by medical evaluation, including medical and psychiatric history, physical and neurological examinations, ECG, vital sign measurements, and laboratory test results, as evaluated by the investigator
* Ability, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements, including the prescribed dosage regimens, scheduled visits, laboratory tests, and other trial procedures

Exclusion Criteria:

* Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus, thyroid disorders), malignancy, hematological, immunological, neurological, or psychiatric disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial
* "Yes" responses for any of the following items on the C-SSRS (within the individual's lifetime):

  * Suicidal Ideation Item 3 (Active Suicidal Ideation With Any Methods [Not Plan] Without Intent to Act)
  * Suicidal Ideation Item 4 (Active Suicidal Ideation With Some Intent to Act, Without Specific Plan)
  * Suicidal Ideation Item 5 (Active Suicidal Ideation With Specific Plan and Intent)
  * Any of the Suicidal Behavior items (Actual Attempt, Interrupted Attempt, Aborted Attempt, or Preparatory Acts/Behavior)
* "Yes" responses for any of the following items on the C-SSRS (within past 12 months):

  * Suicidal Ideation Item 1 (Wish to be Dead)
  * Suicidal Ideation Item 2 (Non-Specific Active Suicidal Thoughts) Serious risk of suicide in the opinion of the investigator is also exclusionary
* Any condition or surgery that could possibly affect drug absorption, including, but not limited to, bowel resections, bariatric weight loss surgery/procedures, gastrectomy, and cholecystectomy
* Positive result for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis B total core antibody, or hepatitis C antibody with detectable viral ribonucleic acid (RNA) levels at screening
* Positive drug screen (including cotinine and tetrahydrocannabinol (THC)) or a positive test for alcohol
* Female participants who are pregnant, breastfeeding, or planning to become pregnant during IMP treatment or within 7 days after the last dose of IMP
* Known allergy or hypersensitivity to the IMP, closely related compounds, or any of their specified ingredients
* Received IMP in a clinical trial of emraclidine

NOTE: Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Emraclidine | Predose and up to 96 hours post dose in each treatment period
Time to Maximum Plasma Concentration (Tmax) of Emraclidine | Predose and up to 96 hours post dose in each treatment period
Area Under the Plasma Concentration-time Curve From Time 0 to the time of Last Quantifiable Concentration (AUC0-t) of Emraclidine | Predose and up to 96 hours post dose in each treatment period
Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUCinf) of Emraclidine | Predose and up to 96 hours post dose in each treatment period

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to approximately 4 months
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Results | Up to approximately 4 months
Number of Participants With Clinically Significant Changes in Vital Sign Values | Up to approximately 4 months
Number of Participants With Clinically Significant Changes in Clinical Laboratory Assessments | Up to approximately 4 months
Number of Participants With Clinically Significant Changes in Physical and Neurological Examination Results | Screening up to checkout (up to approximately 4 months)
Changes in Suicidality as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to approximately 4 months
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Overland Park, Kansas, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No